CLINICAL TRIAL: NCT00791206
Title: Single Blind Randomized Controlled Crossover Trial of the Effects of Remote Preconditioning on the Tissue Metabolism During Exercise and Ischemia
Brief Title: Trial of the Effects of Remote Preconditioning on the Tissue Metabolism During Exercise and Ischemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrew Redington, Head, Heart Centre-Cardiology Division, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1000012859
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Ischemia
Keywords: exercise; ischemia; MRI; MRI spectroscopy; Ischemia preconditioning
MeSH Terms: conditions — Ischemia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Real preconditioning
- 2 (Other)
  Interventions: Procedure: Sham preconditioning

INTERVENTIONS:
Procedure: Real preconditioning — Preconditioning will consist of four 5 minutes cycles of upper limb ischemia interspaced with 5 minutes of reperfusion, using a blood-pressure cuff inflated to a pressure 15 mmHg greater than systolic arterial pressure.
  Arms: 1
Procedure: Sham preconditioning — Preconditioning will consist of four 5 minutes cycles of upper limb ischemia interspaced with 5 minutes of reperfusion, using a blood-pressure cuff inflated to a pressure 10mmHg with the same cycling protocol as the real preconditioning.
  Arms: 2

SUMMARY:
Previously, the preconditioning signaling pathways have been studied on molecular level or in animal model. By using MR spectroscopy and imaging in a dynamic human model of preconditioning, we will have a better understanding how mitochondrial and endothelial function are affected by preconditioning in-vivo.

DETAILED DESCRIPTION:
Ischemic preconditioning is a mechanism that protects tissue against ischemia-reperfusion injury. The protective effect of preconditioning is induced by short periods (1-5 minutes) of non-lethal ischemia to the target tissue, which becomes resistant to a prolonged, otherwise lethal, period of ischemia. Despite its proven potency in experimental models, ischemic preconditioning has not reached widespread clinical application because of the difficulties in applying the stimulus to the target organ (eg Heart, Brain), and even brief ischemia to the target organ can cause dysfunction.

Remote ischemic preconditioning (RIPC) is a more clinically relevant stimulus. It has been shown that preconditioning of one coronary territory induces ischemia protection in other parts of the heart. Subsequently, other studies have shown, in rodent models, that preconditioning of one organ (eg kidney) could induce protection in other organs (eg heart). We recently have confirmed, in a series of animal and human preclinical studies, that this concept can be widened; ultimately showing that four 5-minute episodes of ischemia to the skeletal limb muscles (induced by inflating a standard blood pressure cuff to a level higher than the blood pressure) protects the heart and lungs against ischemia-reperfusion injury in children undergoing cardiac surgery using cardiopulmonary bypass.

The current research is designed to investigate with MRI spectroscopy techonology, the potential physiological mechanisms involved in the protective effects of preconditioning, and the effects of ischemia and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Post-pubescent non-athletes between the ages of >16 and <40 years of age.

Exclusion Criteria:

* Older than 40 year old.
* Younger than 16 year old.
* Major medical condition
* Illness, surgery or medical intervention in the last 48 hours.
* Diabetes Mellitus
* Caffeine intake in the last 48 hours
* Athlete (more than 5 training sessions per week)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in mitochondrial function following the preconditioning as evidenced by a faster rate of recovery of phosphocreatinine after exercise. | 2 hours
Improvement of endothelial and microvascular dysfunction induced by 20 minutes of forearm ischemia. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redington, MD, Principal Investigator — The Hospital for Sick Children